CLINICAL TRIAL: NCT02236819
Title: EuReCa ONE : An International, Prospective, Multi-centre, One Month Survey of Epidemiology, Treatment and Outcome of Patients Suffering an Out-of-hospital Cardiac Arrest in Europe
Brief Title: A Multi-centre Survey of Epidemiology, Treatment and Outcome of Patients Suffering an Out-of-hospital Cardiac Arrest
Acronym: EuReCaONE
Status: Completed | Type: Observational
Sponsor: German Resuscitation Registry (Other)
Collaborators: European Resuscitation Council (ERC) (Unknown)
Responsible Party: Principal Investigator, Jan-Thorsten Graesner, MD, Medical Director Emergency Medicine University Hospital Schleswig-Holstein, Campus Kiel, Germany, German Resuscitation Registry
Other Study IDs: eureca1-2014; eureca 2014 (Other: German Resuscitation Registry)
Record Dates: First submitted 2014-09-02; First posted 2014-09-11 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
There is considerable variation in the incidence of out-of-hospital cardiac arrest (OHCA) across Europe. The likelihood of attempted resuscitation also varies. To better understand the factors that contribute to variation, more data on incidence, management and outcomes from OHCA is required. A European, multi-centre study provides the opportunity to uncover differences throughout Europe and may help find explanations for these differences. Results may also have potential to support the development of quality benchmarking between European Emergency Medical Services (EMS).

This prospective European study will involve 27 different countries. It provides a common Utstein-based dataset, data collection methodology and a common data collection period for all participants, thereby potentially increasing comparability.

Study research questions will address the following: OHCA incidence in different European regions; incidence of cardiopulmonary resuscitation (CPR) attempted; initial presenting rhythm in patients where bystanders or EMS starts CPR or any other resuscitation intervention; rate of any return of spontaneous circulation (ROSC); patient status at handover to a hospital i.e. ROSC, ongoing CPR, dead; incidence of patients still alive 30 days after OHCA; incidence of patients discharged alive from hospital.

DETAILED DESCRIPTION:
The participating registries will transfer unprocessed anonymised data. Transmission of aggregated data should be avoided whenever possible; only in case of limitations due to national laws or ethical requirements should a participating registry transmit aggregated data. Every single case requires a data sheet (DS). Data will be collected within the national, regional or local participating registries (either as a computer-based export from the national, regional or local registry or as a paper-based DS. After validation and anonymisation of data by participating registries the data will then be transferred only via the national coordinator (computer-based) to the study centre. National coordinators are responsible for quality control i.e. the completeness reliability and accuracy of the of data, including timely submission of data to the study management group. Every DS will be identified by a unique number, including the country and region of origin. Registries that cannot transfer unprocessed original data due to the reasons mentioned above will collect data themselves. These registries will then send aggregated data to the study centre. Participating registries must collect basic EMS data on the region and population served. This registry-specific information must only be transmitted once during the study period. Data (computer and paper-based) will be handled according to national laws concerning data security; the national coordinator is responsible for maintaining the necessary standards. Access to the data will be protected by username and password.

ELIGIBILITY:
Inclusion Criteria:

* All patients who suffer an out of hospital cardiac arrest and are attended by the EMS at any stage during the event.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of 27 European countries
Sampling Method: Non-Probability Sample
Enrollment: 10682 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
incidence of patients still alive 30 days after out of hospital cardiac arrest or patients discharged alive from hospital | 30 days after OHCA
  co primary outcome is ROSC/admission to hospital in cases, victims have no ROSC or died on scene

SECONDARY OUTCOMES:
patient status at handover to a hospital | Hospital admission after EMS treatment (within first 24h after OHCA)
  Timepoint/Timestamp within the first 24 hours after EMS treatment started
return of spontaneous circulation | during the time period of EMS treatment within the first 24 h after OHCA
  ROSC at any time during the treatment of EMS after OHCA during the first 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Thorsten Gräsner, MD, Principal Investigator — German Resuscitation Registry
Locations (1):
- Germany ans 26 other european registries, Kiel, Germany

REFERENCES:
- [Background] Grasner JT, Bottiger BW, Bossaert L; European Registry of Cardiac Arrest (EuReCa) ONE Steering Committee; EuReCa ONE Study Management Team. EuReCa ONE - ONE month - ONE Europe - ONE goal. Resuscitation. 2014 Oct;85(10):1307-8. doi: 10.1016/j.resuscitation.2014.08.001. Epub 2014 Aug 15. No abstract available. PMID 25132474
- [Derived] Wnent J, Masterson S, Grasner JT, Bottiger BW, Herlitz J, Koster RW, Rosell Ortiz F, Tjelmeland I, Maurer H, Bossaert L. EuReCa ONE - 27 Nations, ONE Europe, ONE Registry: a prospective observational analysis over one month in 27 resuscitation registries in Europe - the EuReCa ONE study protocol. Scand J Trauma Resusc Emerg Med. 2015 Jan 24;23:7. doi: 10.1186/s13049-015-0093-3. PMID 25927980
- See also: Official study website — http://www.eureca-one.eu